CLINICAL TRIAL: NCT06594965
Title: Phase II Study on the Efficacy, Safety, and Pharmacokinetics of HS-20106 in Patients With IPSS-R Very Low-risk, Low-risk, or Moderate-risk Myelodysplastic Syndrome (MDS) Anemia
Brief Title: A Study of HS-20106 to Treat Anemia Due to Very Low, Low, or Intermediate Risk Myelodysplastic Syndromes
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-20106-201
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Myelodysplastic Syndromes; Anemia; MDS; Bone Marrow Disease
Keywords: MDS; HS-20106; KER-050; fusion protein; TGF-β
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia; Bone Marrow Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HS-20106 Cohort 1 (Experimental): Part A: Non-transfusion dependent population
  Interventions: Drug: HS-20106
- HS-20106 Cohort 2 (Experimental): Part A: Transfusion-Dependent Population（low-transfusion burden (LTB) and high-transfusion burden (HTB)）
  Interventions: Drug: HS-20106

INTERVENTIONS:
Drug: HS-20106 — HS-20106 administered subcutaneously every 4 weeks for up to 6 cycles. Eligible participants may be able to continue to receive subcutaneously administered HS-20106 after completing 6 cycles in the extended treatment period.

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and pharmacokinetics of HS-20106 on anemia in patients with very low, low or intermediate risk MDS.

DETAILED DESCRIPTION:
Anemia is considered to be one of the most prevalent cytopenias in patients who have myelodysplastic syndromes, an umbrella term used to describe disorders relating to the ineffective production of red blood cells, white blood cells, and/or platelets. The goal of this study is to assess the efficacy, safety and PK of HS-20106 on anemia in Chinese patients with very low, low or intermediate risk MDS. Eligible subjects will be treated with HS-20106. Patients should be treated for at least 24 weeks in the core treatment period to assess their response to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MDS according to World Health Organization (WHO) classification that meets Revised International Prognostic Scoring System (IPSS-R) classification of very low, low, or intermediate risk disease（IPSS-R ≤ 3.5）.
2. < 5% blasts in bone marrow and < 1% blasts in peripheral blood.
3. Each cohort is defined as:

   Cohort 1： In NTD participants, having received no red blood cell (RBC) transfusions within 16 weeks Hgb concentration between 60 and 100g/L.

   Cohort 2： In LTB participants, having received an average of < 4 units of RBC transfused within 8 weeks (i.e., total blood transfused over 16 weeks/2) Hgb concentration between 60 and 100 g/L.

   In HTB participants, having received an average of ≥ 4 units of RBC transfused within 8 weeks (i.e., total blood transfused over 16 weeks/2) Hgb concentration between 60 and 100 g/L.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 (if related to anemia.
5. Females of child-bearing potential and sexually active males must agree to use effective methods of contraception.

Exclusion Criteria:

1. Chromosome 5q deletion, del (5q).
2. Anemia caused by other reasons, such as iron deficiency anemia, megaloblastic anemia, aplastic anemia, renal anemia or blood loss.
3. Diagnosis of secondary MDS (i.e., MDS known to have arisen as the result of chemical injury or treatment with chemotherapy and/or radiation for other diseases).
4. Prior treatment with azacitidine, decitabine, lenalidomide, luspatercept, or sotatercept.
5. Treatment within 4 weeks prior to C1D1 with:

1) Erythropoiesis stimulating agent (ESA) OR 2) Granulocyte colony-stimulating factor (G-CSF) OR 3) Granulocyte-macrophage colony-stimulating factor (GM-CSF) 6. Iron chelation therapy if initiated within 8 weeks prior to C1D1. 7. Vitamin B12 therapy if initiated within 8 weeks prior to C1D1. 8. Treatment with another investigational drug or device or approved therapy for investigational use < or = 4 weeks prior to C1D1, or if the half-life of the previous product is known, within 5 times the half-life prior to C1D1, whichever is longer.

9. Peripheral blood white blood cell count >13.0 x 10*9/L. 10. Neutrophil count < 1.0 x 10*9/L. 11. Platelet count > 450 x 10*9/L or < 30 x 10*9/L. 12. Transferrin saturation < 15%. 13. Ferritin < 15 μg/L. 14. Folate < 4.5 nmol/L (< 2.0 ng/mL). 15. Vitamin B12 < 148 pmol/L (< 200 pg/mL). 16. Estimated glomerular filtration rate (GFR) < 40 mL/min/1.73 m2 (as determined by the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI].

17. Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who achieve modified 2006 International Working Group (IWG)Hematologic Improvement-Erythroid (HI-E) response | Week 1 through Week 24
  * In NTD and LTB participants, response is defined as a mean hemoglobin (Hgb) increase of ≥ 15 g/L from Baseline during any consecutive 8-week period during the treatment period (in the absence of RBC transfusions)
  * In HTB participants, response is defined as a reduction by ≥ 4 units of RBCs transfused during any consecutive 8-week period on study compared with Baseline

SECONDARY OUTCOMES:
HI-E Duration | Throughout the study period, assessed up to 48 weeks.
  the maximum duration of meeting the HI-E criteria for a subject who achieved HI-E.
Time to HI-E | Week 1 through Week 24
  the time from the first dose of study drug to the first achievement of HI-E.
Proportion of participants with RBC-TI ≥ 8 Weeks（cohort 2 only） | Week 1 through Week 24
  the proportion of participants who did not require RBC transfusion for at least 1 consecutive 8-week period.
Duration of TI response | Throughout the study period, assessed up to 48 weeks.
  the longest duration of response for participants who achieved RBC-TI of ≥ 8 weeks during the treatment period
Time to RBC-TI ≥ 8 weeks | Week 1 through Week 24
  the time from the first dose of study drug to the first achievement of RBC-TI ≥ 8 weeks.
The proportion of participants with progression to intermediate-risk (IPSS-R score > 3.5) and higher MDS or AML. | Week 1 through Week 24
  Percentage of participants progressing to intermediate-risk (IPSS-R score > 3.5) or higher MDS or AML throughout the course of the study
Time to progression to intermediate-risk (IPSS-R score > 3.5) or higher MDS or AML. | Week 1 through Week 24
  Time to progression was defined as the time between the first dose date and the first diagnosis of progression.
Incidence of adverse events (AEs) and serious adverse events (SAEs). | Throughout the study period, assessed up to 48 weeks.
  Type, frequency, severity of AEs and relationship of AEs to HS-20106
Pharmacokinetic- AUC | Throughout the study period, assessed up to 48 weeks.
  Pharmacokinetics of HS-20106
Pharmacokinetic- Cmax | Throughout the study period, assessed up to 48 weeks.
  Maximum plasma concentration of drug
Antidrug antibodies (ADA) | Throughout the study period, assessed up to 48 weeks.
  Frequency of antidrug antibodies and effects on efficacy, safety or PK

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Blood Diseases Hospital, Tianjin, Tianjin Municipality, China